CLINICAL TRIAL: NCT03761745
Title: Rotational Stability of Different Intraocular Lenses in The Capsular Bag
Status: Completed | Type: Observational
Sponsor: Wenzhou Medical University (Other)
Responsible Party: Principal Investigator, A-Yong Yu, Rotational Stability of Different Intraocular Lenses in The Capsular Bag, Wenzhou Medical University
Other Study IDs: 2018Rotation
Record Dates: First submitted 2018-11-26; First posted 2018-12-03 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Intraocular Lens Complication; Phacoemulsification
Keywords: Rotation; Postoperative Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To evaluate the rotational stability difference among different intraocular lens. The rotational stability is evaluated by measurement of rotation of the IOL after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Patients who had received Femtosecond laser-assisted phacoemulsification surgery with IntelliAxis-L capsular mark.
* The operation was smooth and there were no surgical complications.

Exclusion Criteria:

* Corneal and other ocular diseases (such as corneal opacity, keratitis, glaucoma, uveitis, lens dislocation or subluxation, lens capsule relaxation, retinopathy, etc.);
* History of ocular trauma or surgery before this cataract surgery;
* intraoperative and postoperative complications, such as posterior capsule rupture, corneal endothelium decompensation;
* Patients with severe or unstable heart, liver, kidney, lung, endocrine (including thyroid dysfunction), blood, mental dysfunction and other diseases affect the results of this study;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who received Femtosecond laser-assisted phacoemulsification surgery in The Eye Hospital of Wenzhou Medical University
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2018-12-29 (Actual); Primary Completion 2024-10-30 (Actual); Study Completion 2024-10-30 (Actual)

PRIMARY OUTCOMES:
Alignment of intraocular lens | 1 day postoperatively
  The alignment of intraocular lens was evaluated by anterior segment photography
Alignment of intraocular lens | 1 week postoperatively
  The alignment of intraocular lens was evaluated by anterior segment photography
Alignment of intraocular lens | 1 month, postoperatively
  The alignment of intraocular lens was evaluated by anterior segment photography

SECONDARY OUTCOMES:
Intraocular Pressure | 1 day, 1 week, 1 month, postoperatively
  Intraocular Pressure measured by non-contact tonometers
Corrected Visual Acuity (UCVA) at Distance | 1 day, 1 week, 1 month, postoperatively
  UCVA was determined by subjective refraction
Uncorrected Visual Acuity (UCVA) at Distance | 1 day, 1 week, 1 month, postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: AYong Yu, MD.PhD., Principal Investigator — Wenzhou Medical University
Locations (1):
- Eye Hispital of Wenzhou Medical University, Wenzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No